CLINICAL TRIAL: NCT02954523
Title: Phase I/II Study of Dasatinib and Osimertinib (AZD9291) in Patients With Advanced Non-small Cell Lung Cancer With EGFR Mutations
Brief Title: Dasatinib and Osimertinib (AZD9291) in Advanced Non-Small Cell Lung Cancer With EGFR Mutations
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Chul Kim (Other)
Collaborators: AstraZeneca (Industry); Bristol-Myers Squibb (Industry); Walter Reed National Military Medical Center (U.S. Federal Agency); Hackensack Meridian Health (Other)
Responsible Party: Sponsor-Investigator, Chul Kim, Assistant Professor, Georgetown University
Organization: Georgetown University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0493
Record Dates: First submitted 2016-10-25; First posted 2016-11-03 (Estimated); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: EGFR Gene Mutation; Nonsmall Cell Lung Cancer
Keywords: NSCLC; Non-small cell; Lung Cancer; Dasatinib; Osimertinib; AZD9291; EGFR Mutations; Epidermal growth factor receptor (EGFR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Dasatinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase I- Dasatanib Dose Level 1 (Experimental): Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at up to 4 dose levels. Level 1 (the starting dose - 50 mg twice daily).
  Dose escalation will only include 2 dose levels (Levels 1 and 2); in addition there will be 2 dose levels below the starting dose level if dose reductions are necessary (Levels -1 and -2).
  There is no limit to the number of cycles a patient can receive.
  Interventions: Drug: Dasatinib; Drug: Osimertinib
- Phase I- Dasatanib Dose Level 2 (Experimental): Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at up to 4 dose levels. Level 2 (70 mg twice daily).
  Dose escalation will only include 2 dose levels (Levels 1 and 2); in addition there will be 2 dose levels below the starting dose level if dose reductions are necessary (Levels -1 and -2).
  There is no limit to the number of cycles a patient can receive.
  Interventions: Drug: Dasatinib; Drug: Osimertinib
- Phase I- Dasatanib Dose Level -1 (Experimental): Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at up to 4 dose levels. Level -1 (70 mg once daily).
  Dose escalation will only include 2 dose levels (Levels 1 and 2); in addition there will be 2 dose levels below the starting dose level if dose reductions are necessary (Levels -1 and -2).
  There is no limit to the number of cycles a patient can receive.
  Interventions: Drug: Dasatinib; Drug: Osimertinib
- Phase I- Dasatanib Dose Level -2 (Experimental): Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.d
  Dasatinib is taken orally and will be given at up to 4 dose levels. Level -2 (50 mg once daily).
  Dose escalation will only include 2 dose levels (Levels 1 and 2); in addition there will be 2 dose levels below the starting dose level if dose reductions are necessary (Levels -1 and -2).
  There is no limit to the number of cycles a patient can receive.
  Interventions: Drug: Dasatinib; Drug: Osimertinib
- Phase II- Maximum tolerated dose (Experimental): The phase II portion of the study will use the maximum tolerated dose of dasatinib determined in the phase I portion. Osimertinib (AZD9291) will be given at the same 80mg dose as the phase I portion. There is no limit to the number of cycles a patient can receive.
  Interventions: Drug: Dasatinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Dasatinib — oral every day
  Other Names: BMS-354825
Drug: Osimertinib — oral every day
  Other Names: AZD9291

SUMMARY:
This is a study for patients with advanced non-small cell lung cancer with changes to their cancer cells called EGFR mutations. Mutated EGFR is important in the growth of cancer cells. Medical studies have shown that patients with EGFR mutation-positive lung cancer gain more benefit from targeted therapy drugs such as EGFR inhibitors than with standard chemotherapy. However, a significant proportion of patients carrying these sensitizing mutations do not respond well to the first-generation EGFR-TKIs (erlotinib and gefitinib), indicating the existence of intrinsic resistance mechanisms. Moreover, despite initial response to EGFR-TKIs, acquired resistance is inevitable in all patients.

The investigators have recently shown that Cripto-1 overexpression in EGFR mutant NSCLC contributes to the intrinsic resistance to EGFR-TKIs through activation of the SRC oncogene. They have also shown that a combination of an EGFR-TKI (both erlotinib and osimertinib) and a Src inhibitor are synergistic in Cripto-1 overexpressing tumors in the laboratory.

This study will be testing a combination of two drugs, dasatinib and osimertinib, to overcome resistance to EGFR-TKIs. Osimertinib (AZD9291) is a third-generation EGFR-TKI, which selectively blocks the activity of EGFR mutants, but spares that of wild type. The advantage of using osimertinib is that it inhibits not only the sensitizing EGFR mutations, but also the T790M mutant, which is the most common mechanism of acquired resistance. Dasatinib is a potent, orally available ABL1/SRC TKI, approved for the treatment of chronic myeloid leukemia (CML) in first-line and in patients with imatinib-resistant disease or intolerant, and is being actively studied in patients with advanced solid tumors.

The first part of the study will involve finding the highest dose of dasatinib that can be given with osimertinib without causing severe side effects, finding out the side effects seen by giving dasatinib at different dose levels with osimertinib, and measuring the levels of dasatinib and osimertinib in blood at different dose levels. The second part will determine the effects of the combination of dasatinib and osimertinib and determine if the amount of Cripto-1 protein in your tumor or blood makes you more likely to have a good response to the combination of dasatinib and osimertinib.

DETAILED DESCRIPTION:
The treatment of patients with advanced non-small cell lung cancer is unsatisfactory. The median survival is approximately 12 months with standard chemotherapy. Epidermal growth factor receptor (EGFR) mutations are one of the most frequent genetic abnormalities observed in non-small cell lung cancer (NSCLC), especially in adenocarcinoma subtype. The most predominant EGFR mutations are in-frame deletions in exon-19 and L858R missense mutation, and patients carrying these mutations are mostly sensitive to the EGFR-targeted tyrosine kinase inhibitors (TKIs). However, a significant proportion of patients carrying these sensitizing mutations do not respond well to the first generation EGFR-TKIs (erlotinib and gefitinib), indicating the existence of intrinsic resistance mechanisms. Moreover, despite initial response to EGFR-TKIs, acquired resistance is inevitable in all patients. Novel treatment strategies need to be developed to overcome resistance to EGFR-TKIs. The investigators have recently shown that Cripto-1 overexpression in EGFR mutant NSCLC contributes to the intrinsic resistance to EGFR-TKIs through SRC activation. They have also shown that a combination of an EGFR-TKI (both erlotinib and AZD9291) and a Src inhibitor are synergistic in vitro and in vivo in Cripto-1 overexpressing tumors. AZD9291 is a third-generation EGFR-TKI, which selectively blocks the activity of EGFR mutants but spares that of wild type. The advantage of using AZD9291 is that it inhibits not only the mutants of exon-19 deletion and L858R, but also the T790M mutant, which is the most common mechanism of acquired resistance. Dasatinib is a potent, orally available ABL1/SRC TKI, approved for the treatment of chronic myeloid leukemia (CML) in first-line and in patients with imatinib-resistant disease or intolerant, and is being actively studied in patients with advanced solid tumors.

This is an open-label, non-randomized, prospective phase I/II trial. The phase I portion will follow a standard 3+3 design for the phase I portion and one-sample group sequential multiple testing procedure for the phase II portion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically or histologically confirmed advanced NSCLC. Patients with mixed histology containing a small cell lung cancer component are not eligible.
* Patients must have adequate archival material from a previous biopsy to determine EGFR mutation status and Cripto-1 expression, or undergo a biopsy of fresh tissue of the primary cancer or a metastatic site in order to make these determinations, if archival material is not available.
* Presence of sensitizing EGFR mutations (deletion in exon 19, L858R in exon 21, G719X, and L861Q). Patients with the T790M mutation will also be eligible.
* No prior treatment with an EGFR TKI for the advanced NSCLC.
* ECOG performance status of 0-2.
* Patients must have measurable disease by RECIST criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 7.1.2 for the evaluation of measurable disease.
* Prior systemic treatment is allowed, but toxicities of prior therapy must be resolved to grade 1 or less as per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
* Adequate organ and bone marrow function (hemoglobin > 9 g/dL; absolute neutrophil count > 1.5 x 109/L; platelet counts > 100 x 109/L; serum bilirubin < 2 x ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN or < 5 x ULN if liver metastases; calculated creatinine clearance > 50 mL/min).
* No uncontrolled arrhythmia; no myocardial infarction in the last 6 months.
* Life expectancy of at least 12 weeks.
* Age > 18 years.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had radiotherapy (except for palliative reasons), immunotherapy or chemotherapy during the previous 4 weeks (6 weeks for nitrosoureas or mitomycin) before treatment, or those who have ongoing toxic manifestations of previous treatments, with the exception of alopecia, of grade higher than 1.
* Major thoracic or abdominal surgery from which the patient has not sufficiently recovered yet.
* Untreated and uncontrolled second tumor in the past 2 years.
* Logistical or psychological hindrance to participation in clinical research.
* Patients with untreated symptomatic brain metastases may be eligible if symptoms do not require urgent surgery or radiation, and no steroids are necessary.
* Patients with evidence of interstitial lung disease (bilateral, diffuse, parenchymal lung disease).
* Pleural or pericardial effusions of any grade at study entry. Subjects previously diagnosed with pleural/pericardial effusion of any grade resolved at the time of study entry are allowed.
* Ability to become pregnant (or already pregnant or lactating). Women and men who want to participate have to agree to use two highly effective forms of contraceptive prior to study entry, for the duration of study participation, and for 30 days following completion of therapy, to be eligible. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
* At high medical risk because of non-malignant systemic disease including uncontrolled infection.
* Known to be serologically positive for hepatitis B, hepatitis C or HIV.
* Uncontrolled or significant cardiovascular disease, including any of the following:

  * QTc interval > 480 msec (mean value and manually verified) at 3 or more time points within a 24 hour period if necessary.
  * Diagnosed or expected congenital long QT syndrome.
  * Concurrent congestive heart failure, prior history of class III/IV cardiac disease (New York Heart Association).
  * Left ventricular ejection fraction < 50%
  * Prior history of cardiac ischemia or cardiac arrhythmia within the last 6 months. Coronary angioplasty or stenting in the previous 12 months.
  * Any history of second or third degree heart block (may be eligible if the subject currently has a pacemaker).
  * Uncontrolled hypertension defined as inability to maintain blood pressure below the limit of 140/90 mmHg.
  * Known pulmonary hypertension.
* History of significant bleeding disorder unrelated to CML, including:

  * Diagnosed congenital bleeding disorders (e.g. von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g. acquired anti-factor VII antibodies)
* Any other medical condition that in the Investigator's opinion would not make the patient a good candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD PhD, Study Chair — Associate Director for Clinical Research, Lombardi Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cacner Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim C, Liu SV, Crawford J, Torres T, Chen V, Thompson J, Tan M, Esposito G, Subramaniam DS, Giaccone G. A Phase I Trial of Dasatinib and Osimertinib in TKI Naive Patients With Advanced EGFR-Mutant Non-Small-Cell Lung Cancer. Front Oncol. 2021 Sep 8;11:728155. doi: 10.3389/fonc.2021.728155. eCollection 2021. PMID 34568058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study accrual terminated early and no subjects enrolled into the phase II portion of the study.
Groups:
- Phase IPhase I- Dasatinib Dose Level 2: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule. Dasatinib is taken orally Level 2 (70mg twice daily). There is no limit to the number of cycles a patient can receive.
- Phase 1- DasatinibDose Level 1: Osimertinib(AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule. Dasatinib is taken orally Level 1 (50mg twice daily). There is no limit to the number of cycles a patient can receive.
- Phase 1- DasatinibDose Level -1: Osimertinib (AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule. Dasatinib is taken orally Level -1 (70mg once daily). There is no limit to the number of cycles a patient can receive.
Period: Overall Study
Arm/Group | Phase IPhase I- Dasatinib Dose Level 2 | Phase 1- DasatinibDose Level 1 | Phase 1- DasatinibDose Level -1
Started | 3 | 6 | 1
Completed | 3 | 6 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I- Dasatinib Dose Level 2: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level 2 (70 mg twice daily).
- Phase 1- Dasatinib Dose Level 1: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level 1 (50 mg twice daily).
- Phase 1- Dasatinib Dose Level -1: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level -1 (70 mg once daily),
- Total: Total of all reporting groups
Arm/Group | Phase I- Dasatinib Dose Level 2 | Phase 1- Dasatinib Dose Level 1 | Phase 1- Dasatinib Dose Level -1 | Total
Number analyzed (Participants) | 3 | 6 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 0 | 3
  >=65 years | 1 | 5 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 1 | 9
  Male | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 3 | 1 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I : Number of Patients With Drug-related Adverse Events as Assessed by CTCAEv4.0
Description: Number of patients with drug related adverse events (Dose Limiting Toxicities) on dasatinib when given in combination with osimertinib
Time Frame: Cycle 1 (28 day cycle)
Measure: Number; unit: participants
Groups:
- Phase I- Dasatinib Dose Level 2: Osimertinib (AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level 2 (70 mg twice daily).
- Phase 1- Dasatinib Dose Level 1: Osimertinib (AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level 1 (50 mg twice daily).
- Phase 1- Dasatinib Dose Level -1: Osimertinib (AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level -1 (70 mg once daily),
Arm/Group | Phase I- Dasatinib Dose Level 2 | Phase 1- Dasatinib Dose Level 1 | Phase 1- Dasatinib Dose Level -1
Number analyzed (Participants) | 3 | 6 | 1
participants | 0 | 3 | 0

2. Primary Outcome: Phase II : Number of Patients That do Not Progress According to RECIST v1.1
Description: The rate of patients non-responding (progressive disease or stable disease lasting 4 months or less) to the combination of osimertinib and dasatinib
Time Frame: 9 months
Population: Study close to accrual early. No participants enrolled in phase II.
Groups:
- Phase II: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at up to 4 dose levels. Level -2 (50 mg once daily), Level -1 (70 mg once daily), Level 1 (the starting dose - 50 mg twice daily), Level 2 (70 mg twice daily).
  Dose escalation will only include 2 dose levels (Levels 1 and 2); in addition there will be 2 dose levels below the starting dose level if dose reductions are necessary (Levels -1 and -2).
  There is no limit to the number of cycles a patient can receive.
  The phase II portion of the study will use the maximum tolerated dose of dasatinib determined in the phase I portion. Osimertinib (AZD9291) will be given at the same 80mg dose as the phase I portion.
  Dasatinib: oral every day
  Osimertinib: oral every day
Arm/Group | Phase II
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With Treatment-related Adverse Events in the Phase II Study
Description: Number of patients with treatment-related adverse events in the phase II study, who are treated at the same dose that has been selected based on the phase I part
Time Frame: 18 months
Population: Study close to accrual early. No participants enrolled in phase II.
Arm/Group | Phase II
Number analyzed (Participants) | 0

4. Secondary Outcome: Concentration of Osimertinib in Blood (Cmax)
Description: To describe the concentration of osimertinib when administered with dasatinib. Blood is obtained from patients before each cycle and 4 hours after start of the first 2 cycles.
Time Frame: 0 hour, 4 hours post dose
Population: Study Terminated early due to lack of enrollment.
Measure: Mean (Full Range); unit: nM/mL
Groups:
- Phase I- Dose Level 1: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at Level 1 (the starting dose - 50 mg twice daily)
  There is no limit to the number of cycles a patient can receive.
  The phase II portion of the study will use the maximum tolerated dose of dasatinib determined in the phase I portion. Osimertinib (AZD9291) will be given at the same 80mg dose as the phase I portion.
  Dasatinib: oral every day Osimertinib: oral every day
- Phase 1- Dose Level 2: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at Level 2 (70 mg twice daily).
  There is no limit to the number of cycles a patient can receive.
  Dasatinib: oral every day Osimertinib: oral every day
- Phase 1- Dose Level -1: Osimertinib (AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level -1 (70 mg once daily),
Arm/Group | Phase I- Dose Level 1 | Phase 1- Dose Level 2 | Phase 1- Dose Level -1
Number analyzed (Participants) | 6 | 3 | 1
nM/mL | 211.5 [166 to 314] | 355 [345 to 365] | 107 [107 to 107]

5. Secondary Outcome: Progression-free Survival
Description: Determination of the time between the start of the experimental treatment and progression of the tumor
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Groups:
- Phase I- Dose Level 2: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at Level 2 (70 mg twice daily). There is no limit to the number of cycles a patient can receive. Dasatinib: oral every day Osimertinib: oral every day
- Phase I- Dose Level -1: Osimertinib (AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level -1 (70 mg once daily),
Arm/Group | Phase I- Dose Level 1 | Phase I- Dose Level 2 | Phase I- Dose Level -1
Number analyzed (Participants) | 6 | 3 | 1
months | 24.7 [3.7 to 31.3] | 10.1 [4.5 to 16.7] | 10.5 [10.5 to 10.5]

6. Secondary Outcome: Overall Survival
Description: From the date of start of the experimental treatment until the date of death from any cause, whichever came first, assessed up to 47 months.
Time Frame: 47 months
Measure: Median (Full Range); unit: months
Groups:
- Dose Level 1: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at Level 1 (the starting dose - 50 mg twice daily) There is no limit to the number of cycles a patient can receive. The phase II portion of the study will use the maximum tolerated dose of dasatinib determined in the phase I portion. Osimertinib (AZD9291) will be given at the same 80mg dose as the phase I portion.
  Dasatinib: oral every day Osimertinib: oral every day
Arm/Group | Dose Level 1 | Phase I- Dose Level 2 | Phase I- Dose Level -1
Number analyzed (Participants) | 6 | 3 | 1
months | 36.1 [23.5 to 46.6] | 16.9 [7.4 to 36.6] | 28.7 [28.7 to 28.7]

7. Secondary Outcome: Duration of Response
Description: Determination of the duration of the response to the treatment, calculated from start of treatment in case of partial response and from the declaration of complete response in case of complete response. The end of the response will be when the tumor progresses
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Groups:
- Phase 1 - Dose Level -1: Osimertinib (AZD9291) will begiven at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally Level -1 (70 mg once daily),
Arm/Group | Phase I- Dose Level 1 | Phase I- Dose Level 2 | Phase 1 - Dose Level -1
Number analyzed (Participants) | 6 | 3 | 1
months | 27.8 [18.6 to 31.9] | 12.2 [8.4 to 15.9] | 8.7 [8.7 to 8.7]

ADVERSE EVENTS:
Time Frame: Up to 6 years.
Description: Study Terminated early due to lack of enrollment. All subjects were analyzed together due to low accrual (too few people in each dose level).
Groups:
- Phase I- Dose Level 1: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at Level 1 (the starting dose - 50 mg twice daily), There is no limit to the number of cycles a patient can receive. Dasatinib: oral every day Osimertinib: oral every day
- Phase I- Dose Level -1: Osimertinib (AZD9291) will be given at a 80mg/day dose taken orally across all levels of the dose escalation schedule.
  Dasatinib is taken orally and will be given at Level -1 (70 mg once daily). There is no limit to the number of cycles a patient can receive.
  Dasatinib: oral every day Osimertinib: oral every day
Arm/Group | Phase I- Dose Level 1 | Phase I- Dose Level 2 | Phase I- Dose Level -1
All-Cause Mortality (participants affected / at risk) | 1/6 | 2/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I- Dose Level 1 (N=6) | Phase I- Dose Level 2 (N=3) | Phase I- Dose Level -1 (N=1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | NA — Worsening Atrial Fibrillation, symptomatic
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | NA
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | NA
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | NA — aphasia
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | NA — central nervous system necrosis due to radiation
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | NA
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Lung infection (Infections and infestations) | 1 (2) | 0 (0) | NA
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | NA — toe infection
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | NA
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | NA
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1) | NA — Right Leg Deep Venous Thrombosis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I- Dose Level 1 (N=6) | Phase I- Dose Level 2 (N=3) | Phase I- Dose Level -1 (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 (2) | 0
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (7) | 2 (3) | 1 (4)
Allergic reaction (Immune system disorders) | 1 (1) | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0
Anemia (Blood and lymphatic system disorders) | 3 (7) | 2 (9) | 0
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 0 | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0
Aspartate aminotransferase increased (Investigations) | 4 (8) | 2 (2) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Bronchial infection (Infections and infestations) | 1 (1) | 0 | 0
Chest Pressure (General disorders) | 1 (2) | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0
Chills (General disorders) | 0 | 1 (1) | 0
Conjunctivitis (Eye disorders) | 2 (2) | 0 | 0
Constipation (Gastrointestinal disorders) | 2 (2) | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 0
Creatinine increased (Investigations) | 2 (8) | 0 | 0
Dental caries (General disorders) | 1 (2) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 6 (8) | 3 (3) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Dysgeusia (Nervous system disorders) | 2 (2) | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (8) | 0
Edema face (General disorders) | 1 (1) | 1 (2) | 0
Edema limbs (General disorders) | 1 (1) | 1 (2) | 0
Ejection fraction decreased (Investigations) | 1 (1) | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 3 (6) | 1 (2) | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 | 0 — Eye Hemmorhage
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 | 0 — tearing of eyes
Fatigue (General disorders) | 4 (14) | 1 (1) | 0
Fever (General disorders) | 3 (5) | 2 (4) | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0
Headache (Nervous system disorders) | 3 (4) | 0 | 0
Heartburn (General disorders) | 1 (1) | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4) | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 | 0 — Covid19
Insomnia (Psychiatric disorders) | 0 | 1 (2) | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0
Mucosal infection (Infections and infestations) | 1 (1) | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 | 0
Nail infection (Infections and infestations) | 1 (1) | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (2) | 1 (3)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (30) | 2 (4) | 1 (2)
Pain (General disorders) | 1 (1) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 | 0
Palpitations (Cardiac disorders) | 2 (3) | 0 | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 (2) | 0
Paronychia (Infections and infestations) | 3 (4) | 0 | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Platelet count decreased (Investigations) | 4 (9) | 1 (2) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (4) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 (3) | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Seizure (Nervous system disorders) | 1 (1) | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 — skin rash
Skin infection (Skin and subcutaneous tissue disorders) | 1 (3) | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 (2) | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 (1) | 0 — Right Leg Deep Venous Thrombosis
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 (11) | 0 — Arteriovenous malformation (AVM)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 0
Watering eyes (Eye disorders) | 1 (1) | 0 | 0
Weight gain (Investigations) | 1 (1) | 0 | 0
Weight loss (Investigations) | 1 (2) | 0 | 1 (2)
White blood cell decreased (Investigations) | 1 (3) | 2 (3) | 1 (4)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 | 0
Urinary tract infection (Infections and infestations) | 1 (1) | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT02954523/Prot_SAP_000.pdf